CLINICAL TRIAL: NCT02778542
Title: Bidirectional Text Messaging for Measurement and Motivation of Medication Adherence in Hypertension, a Pilot Study
Acronym: Way2Text
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 824815
Record Dates: First submitted 2016-05-12; First posted 2016-05-20 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Hypertension
Keywords: Automated Hovering; Remote Monitoring; Bidirectional Text Messaging
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Care Provider, Investigator

ARMS (3):
- Electronic Pill Bottle (Active Comparator): Participants will be mailed an electronic pill bottle for their blood pressure medication.These pill bottles will track how often the participant opens the bottle to take their medication and will transmit that information to study team via cellular data. Participants will also receive a daily text message reminder to take your blood pressure medication.
  Interventions: Behavioral: Electronic Pill Bottle
- Bidirectional Text Messaging (Active Comparator): Participants assigned to bi-directional texting, will receive a daily text message reminder to take their blood pressure medication. Patients in this arm are expected to send a response to the reminder message, indicating if they took their medication that day.
  Interventions: Behavioral: Bidirectional Text Messaging
- Usual Care (No Intervention): Participants in this arm do not receive a medication reminder system.

INTERVENTIONS:
Behavioral: Electronic Pill Bottle — Patients receive electronic pill bottle for their blood pressure medication. Study team can monitor pill bottle openings. Patients also receive daily text reminders to take their blood pressure medication.
  Arms: Electronic Pill Bottle
Behavioral: Bidirectional Text Messaging — Patients receive daily text reminders to take their blood pressure medication. Patients are asked to text their adherence daily.
  Arms: Bidirectional Text Messaging

SUMMARY:
The goal of this pilot study is to test different approaches to monitor medication adherence in hypertension patients, leveraging the NIH-funded Way to Health platform. Patients with poor blood pressure control will be recruited from the University of Pennsylvania Health System practices and offered remote monitoring with electronic pill bottles, bidirectional text messaging or usual care. Our aim is to analyze and compare the effects of remote monitoring with electronic pill bottles versus bidirectional messaging on blood pressure reduction after 4 months.

DETAILED DESCRIPTION:
The goal of this pilot study is to test different approaches to monitor medication adherence in hypertension patients, leveraging the NIH-funded Way to Health platform. Patients with poor blood pressure control will be recruited from the University of Pennsylvania Health System and offered remote monitoring with electronic pill bottles or bidirectional text messaging. Our aim is to analyze and compare the effects of remote monitoring with electronic pill bottles versus bidirectional messaging on blood pressure reduction after 4 months.

Patients will be randomized 2:2:1 to Arm A (electronic pill bottle), Arm B (bidirectional messaging), and Arm C (usual care). A total of 150 participants will be enrolled in the study, with 60 in each intervention arm and 30 in the control. After 4 months all patients will complete an in-person follow-up blood pressure measurement and end of program survey. We will monitor all patient's medical records for an additional 8 months after the intervention to track blood pressure measurement and number of outpatient visits.

Accrual: Participants in this study will be patients being treated within the UPHS health system. They will be identified via daily electronic medical records review by our study staff. The study staff will work with UPHS to create a filter for the electronic medical record system that will generate a monthly list of patients who may meet the study criteria. A study coordinator will review the list of patients to determine eligibility. If patients meet the minimal requirements they will be added to the study screening data base and contacted via recruitment letter and up to 3 follow-up phone calls. The intervention of the study will be 4 months from date of consent, and an additional 8 months of follow-up, passively monitoring visit utilization and blood pressure in the electronic medical record. After a patient enrolls a message will be sent to their PCP via EPIC to notify their physician that their patient is enrolled in our study. At the conclusion of the intervention, participants will complete an in-person blood pressure measurement and post-study survey. Information about BP measurements will be recorded in EPIC and message will be sent to the PCP with the research BP measurement included.

Analysis Plan: The primary outcome will be the systolic blood pressure during the 4 month visit, controlling for the initial systolic blood pressure. Additional outcomes include, percent that are normotensive, recruitment and attrition rates, and patient perceptions about intervention from survey. We will also track BP measurements from the EMR that is obtained through usual care as well as utilization of PCP visits, MPM messaging, and phone calls. We will also compare medication adherence between patients with the electron pill bottles and the patients with bidirectional messaging. Assuming 5.3mmHg standard deviation of SBP (given variability of BP over time) and a two-sided significance level of 0.017 (to accommodate the three pairwise comparisons), our sample size of 60 in each intervention arm and 30 in the control arm provides 80% power to detect a difference in SBP reduction of 3.75 mmHg between either intervention and usual care, and a difference in SBP reduction of 3.1 mmHg between the electronic pill bottle and bidirectional text messaging arms.

Data Safety: Paper-based records will be kept in a secure location and only be accessible to personnel involved in the study. Computer-based files will only be made available to personnel involved in the study through the use of access privileges and passwords.

Prior to access to any study-related information, personnel will be required to sign statements agreeing to protect the security and confidentiality of identifiable information.

Wherever feasible, identifiers will be removed from study-related information. Precautions are in place to ensure the data is secure by using passwords and encryption, because the research involves web-based surveys.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension patients aged 18-75
* At least two clinic visits in the past 12 months
* Blood pressure readings in the last two visits that exceed recommended guidelines (150/90 or 140/90 if aged 21-59 yrs. or with diabetes or nondiabetic CKD).
* Cellular phone with text messaging capabilities
* Prescribed at least one medication for hypertension

Exclusion Criteria:

* Will not or cannot give consent
* Diagnosed with dementia, end stage renal disease, cirrhosis, or metastatic cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | after 4 month intervention
  The primary outcome will be the systolic blood pressure during the 4 month in-person visit, controlling for the initial systolic blood pressure

SECONDARY OUTCOMES:
Medication Adherence | 4 month intervention
  We will compare medication adherence between patients with the electronic pill bottles and the patients with bidirectional messaging.
Passive EMR monitoring | 12 months, including 4 months of intervention and 8 months after intervention
  We will also track BP measurements from the EMR that is obtained through usual care as well as utilization of PCP visits, MPM messaging, and phone calls.

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania

REFERENCES:
- [Derived] Mehta SJ, Volpp KG, Troxel AB, Day SC, Lim R, Marcus N, Norton L, Anderson S, Asch DA. Electronic Pill Bottles or Bidirectional Text Messaging to Improve Hypertension Medication Adherence (Way 2 Text): a Randomized Clinical Trial. J Gen Intern Med. 2019 Nov;34(11):2397-2404. doi: 10.1007/s11606-019-05241-x. Epub 2019 Aug 8. PMID 31396815